CLINICAL TRIAL: NCT00249847
Title: A Feasibility Study of Positron Emission Tomography (PET) of the Serotonin Transporter (SERT) Before and After Treatment With Conjugated Equine Estrogen or Paroxetine for Hot Flashes
Brief Title: Study of PET Scans and Serotonin in Hot Flashes Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to complete accrual; elected to close the study in April 2008.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKCCC J0360
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-10

CONDITIONS: Hot Flashes
Keywords: Hot flashes, vasomotor symptoms, estrogen, paroxetine
MeSH Terms: conditions — Hot Flashes | interventions — Paroxetine; Estrogens, Conjugated (USP)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paroxetine (Experimental): Paroxetine controlled-release (2-12.5 mg tablets, orally, every day for 4 weeks)
  Interventions: Drug: Paroxetine controlled-release
- Conjugated equine estrogen (Experimental): Conjugated equine estrogen (0.625 mg tablet, orally, every day for 4 weeks)
  Interventions: Drug: Conjugated equine estrogen

INTERVENTIONS:
Drug: Paroxetine controlled-release — 2-12.5 mg tablets, orally, every day for 4 weeks
  Other Names: Paxil CR
  Arms: Paroxetine
Drug: Conjugated equine estrogen — 0.625 mg tablet, orally, every day for 4 weeks
  Other Names: Premarin
  Arms: Conjugated equine estrogen

SUMMARY:
The purpose of this study is to determine in a preliminary manner whether successful therapy of hot flashes can be associated with changes in the serotonin transporter in the brain. The serotonin transporter is important in delivering serotonin into certain portions of the brains (serotonin is a chemical that is important in the control of body temperature, mood, sleep, and other functions).

DETAILED DESCRIPTION:
Hot flashes represent the most common complaint among peri- and postmenopausal women. Over 60% of postmenopausal women experience hot flashes, and 10-20% of all postmenopausal women find them nearly intolerable. Despite the prevalence of hot flashes, their pathophysiology is not well understood. Treatment options include non-pharmacological approaches, hormonal interventions, and non-hormonal pharmacological agents. The most effective treatment for hot flashes is estrogen. The most promising non-hormonal treatments for hot flashes are selective serotonin or noradrenergic reuptake inhibitors (SSRI/SNRI). Although estrogen withdrawal is implicated in the initiation of hot flashes, and serotonin's role is well established in thermoregulation, the relationship between estrogen and serotonin is not known. Preclinical studies suggest that both estrogen and SSRI down regulate the serotonin transporter. Clinical studies that further delineate the relationship between effective treatments for hot flashes and the serotonin transporter may shed a new light into the pathophysiology of these symptoms and more importantly, into design of new-targeted treatments.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* 7 or more hot flashes per day for at least 3 months
* Must be able to undergo magnetic resonance (MR) and PET imaging
* Must be able to receive either paroxetine or estrogen

Exclusion Criteria:

* No treatment with hormone therapy or other medications that affect estrogen within the past 3 months
* No evidence of a currently active cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-10; Primary Completion 2007-07 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
To estimate the proportion of women who have a 50% or greater reduction in frequency of hot flashes following 4 weeks of paroxetine or conjugated equine estrogen. | Following 4 weeks of study medication
To evaluate baseline and change in binding of the serotonin transporter in postmenopausal women who suffer hot flashes before and after 4 weeks of paroxetine or conjugated equine estrogen using PET. | Following 4 weeks of study medication
To correlate baseline and change in binding of the serotonin transporter using PET with reduction of hot flashes after 4 weeks of conjugated equine estrogen or paroxetine. | Following 4 weeks of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States